CLINICAL TRIAL: NCT05028426
Title: Single-center Retrospective Study on Safety of Total Knee Replacement Surgery Before and After the Implementation of Enhanced Recovery Program
Brief Title: Safety of Total Knee Replacement Surgery Before and After the Implementation of Enhanced Recovery Program
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/P01/266
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Arthroplasty Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Traditional method of care: Patients managed according to the traditional care protocol without an enhanced recovery program
- Some elements of a fast-track program: operative and postoperative techniques were modified according to a fast-track program
  Interventions: Procedure: Enhanced recovery program
- Full enhanced recovery program: Patients were managed in an enhanced recovery program (elements of the previous fast-track program were modified and preoperative education was added)
  Interventions: Procedure: Enhanced recovery program

INTERVENTIONS:
Procedure: Enhanced recovery program — Enhanced recovery programs are a multimodal approach to optimize patients' physiological and psychological states in the preoperative, intraoperative and postoperative care domains.
  Groups: Full enhanced recovery program; Some elements of a fast-track program

SUMMARY:
The objectives are to describe the transition from traditional care to an enhanced recovery program for the management of total knee arthroplasty, and to evaluate the effect on patient outcomes.

DETAILED DESCRIPTION:
Enhanced recovery programs are an organizational evolution in surgical patient management, in which the patient becomes an actor of his or her own recovery. This multimodal approach aims at optimizing patient physiological and psychological states across preoperative, intraoperative and postoperative domains of care.

At la Rochelle hospital, the decision to take the step happened at the end of 2016. It was proposed by a young surgeon that have been trained on this new approach during his studies and who convinced the head of the surgery department of the benefits for the patients, the healthcare workers, and the institution. The transition took place in two stages, first operative and postoperative techniques were modified, and then preoperative education and counselling were added.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on for posterior-stabilized total knee arthroplasty between January 2015 and December 2018
* unilateral arthroplasty
* a known address for mailing the study information letter

Exclusion Criteria:

* revision arthroplasty
* patients who refused to the use of their data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients were classified into three groups according to the type of care management they received: traditional method of care, some elements of a fast-track program during a transition period, and full enhanced recovery program.
Sampling Method: Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivien Fontaine, MD, Study Director — Groupe Hospitalier La Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. Keywords are Arthroplasty, Replacement, Knee, Enhanced Recovery After Surgery. The available version will be the locked database. The database will be made available by the study director upon request up to 15 years after publication. Medical Subject Headings (MESH) terms will be used to describe clinical data.
  Methodology for will be provided in the publication. International standard unit will be used.
Time Frame: Data will be made available with publication (expected at the end of 2021 or beginning of 2022) and up to 15 years after the end of the study.
Access Criteria: The database will be made available by the study director upon request

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Started | 214 | 132 | 109
Completed | 214 | 132 | 109
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program | Total
Number analyzed (Participants) | 214 | 132 | 109 | 455
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 29 | 36 | 133
  >=65 years | 146 | 103 | 73 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 72 (8.9) | 70 (8.5) | 70 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 77 | 66 | 273
  Male | 84 | 55 | 43 | 182
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 214 | 132 | 109 | 455
American Society of Anesthesiology (ASA) score [Count of Participants; unit: Participants] — The ASA score is a subjective assessment of a patient's overall health that is based on five classes (I to V).
  1. Patient is a completely healthy fit patient.
  2. Patient has mild systemic disease.
  3. Patient has severe systemic disease that is not incapacitating.
  4. Patient has incapacitating disease that is a constant threat to life.
  5. A moribund patient who is not expected to live 24 hour with or without surgery.
  Participants
    ASA score = 1 | 29 | 16 | 16 | 61
    ASA score = 2 | 128 | 87 | 67 | 282
    ASA score = 3 | 57 | 29 | 26 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Early Complication
Description: Recorded complications were Bleeding, Deep periprosthetic joint infection, Implant fracture, Instability, Patellofemoral dislocation, Readmission, Reoperation, Revision, Stiffness, Thromboembolic disease, Tibiofemoral dislocation, Vascular injury, Wound complication.
Time Frame: 3 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
Participants | 9 | 16 | 4

2. Secondary Outcome: Number of Patients With Late Complication
Description: as for outcome 1
Time Frame: up to 28 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
Participants | 0 | 5 | 1

3. Secondary Outcome: Length of Hospital Stay
Description: the time between admission for an operation and discharge from the hospital
Time Frame: up to 1 month after surgery
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
days | 9.5 (2.7) | 5.6 (2.4) | 4.9 (2.1)

4. Secondary Outcome: Preoperative Knee Extension
Description: Measure in degree of how much the knee straightens during consultation with surgeon
Time Frame: up to 1 month before surgery
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
degree | 5 (8.2) | 7.4 (7.4) | 4.8 (8.0)

5. Secondary Outcome: Postoperative Knee Extension
Description: Measure in degree of how much the knee straightens during consultation with surgeon
Time Frame: At 3 months after surgery
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
degree | 0.5 (2.1) | 0.7 (2.8) | 0.8 (3.6)

6. Secondary Outcome: Preoperative Knee Flexion
Description: Measure in degree of how much the knee bends during consultation with surgeon
Time Frame: up to 1 month before surgery
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
degree | 106.5 (13.3) | 107.0 (16.9) | 108.3 (15.7)

7. Secondary Outcome: Postoperative Knee Flexion
Description: Measure in degree of how much the knee bends during consultation with surgeon
Time Frame: At 3 months after surgery
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
Number analyzed (Participants) | 214 | 132 | 109
degree | 114.5 (14.9) | 116.6 (14.4) | 112.9 (16.1)

ADVERSE EVENTS:
Time Frame: The post-surgery follow-up consultation took place 1 month after the operation. Depending on the clinical situation, further follow-up consultations took place up to 28 months after surgery.
Arm/Group | Traditional Method of Care | Some Elements of a Fast-track Program | Full Enhanced Recovery Program
All-Cause Mortality (participants affected / at risk) | 6/214 | 1/132 | 2/109
Serious Adverse Events (participants affected / at risk) | 9/214 | 21/132 | 5/109
Other Adverse Events (participants affected / at risk) | 7/214 | 7/132 | 6/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Method of Care (N=214) | Some Elements of a Fast-track Program (N=132) | Full Enhanced Recovery Program (N=109)
Bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
joint infection (Surgical and medical procedures) | 3 (3) | 8 (8) | 1 (1)
Fracture (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Joint instability (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 2 (2) | 7 (7) | 3 (3)
Stiffness (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vascular injury (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
Wound complication (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Method of Care (N=214) | Some Elements of a Fast-track Program (N=132) | Full Enhanced Recovery Program (N=109)
Fall (General disorders) | 1 (1) | 0 (0) | 1 (1)
Hip surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Joint prosthesis loosening (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (5) | 2 (2) | 2 (2)
Haematoma (Surgical and medical procedures) | 0 (0) | 2 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT05028426/Prot_SAP_000.pdf